CLINICAL TRIAL: NCT03103178
Title: Translation Into Spanish of an Interstitial Lung Disease Quality of Life Questionnaire (KBILD)
Brief Title: Spanish Version of the KBILD Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-KBI-2016-47
Record Dates: First submitted 2017-03-23; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of life questionnaire — Measurement of quality of life

SUMMARY:
The purpose of the present study is to advance in the knowledge of quality of life in patients with ILD by translating a ILD quality of life questionnaire.

There are no specific tools validated in Spanish to evaluate the quality of life in patients with ILD, although these measures are useful for an comprensive evaluation of these patients.

Patients with ILD have a significant impact on their health. If we improve our Knowledge of the different domains affected by the disease, and not only in the pathophysiological ones, we will be able to develop tools to improve their management.

ELIGIBILITY:
Inclusion criteria

1. Subjects older than 18 years.
2. Diagnosis of ILD, established according to the consensus documents of the ATS and ERS [1,2].
3. Acceptance of the patient to participate in the study by signing the informed consent after having discussed with the researchers the objectives, risks and potential benefits.

Exclusion criteria

1. Another chronic respiratory disease other than EPID.
2. Psychiatric disorder or limitation of collaboration (including language, socio-cultural problem, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over 18 years of age diagnosed with diffuse interstitial lung disease for which they are being followed up at the respiratory department of the Santa Creu i Sant Pau Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Validation of a specific quality of life questionnaire for patients with ILD | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain